CLINICAL TRIAL: NCT05759988
Title: Cervical Ripening as an Outpatient Method Using the Foley: a Randomized Trial
Brief Title: Cervical Ripening as an Outpatient Method Using the Foley (COMFORT)
Acronym: COMFORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa Levine, Associate Professor, Division of Maternal Fetal Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 851906
Record Dates: First submitted 2023-02-14; First posted 2023-03-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: Foley balloon catheter; Outpatient cervical ripening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Outpatient cervical ripening with Foley (Experimental): Cervical ripening will begin with a Foley balloon in the outpatient setting
  Interventions: Device: Outpatient Foley catheter
- Standard of care Inpatient cervical ripening (No Intervention): Cervical ripening will begin in the inpatient setting with Foley ballooon or other cervical ripening agent

INTERVENTIONS:
Device: Outpatient Foley catheter — Outpatient Foley catheter placement for induction of labor
  Arms: Outpatient cervical ripening with Foley

SUMMARY:
A multicenter pragmatic randomized trial of nulliparous women undergoing a term (≥37 weeks) induction of labor wherein the provider intends to use a Foley catheter for cervical ripening. The investigators will be comparing outpatient cervical ripening with a Foley catheter to routine inpatient cervical ripening (Foley +/- other method). With this trial, the investigators aim to test our central hypothesis that outpatient Foley will decrease the primary Cesarean Delivery (CD) rate and risk of maternal/neonatal morbidity compared with inpatient cervical ripening.

ELIGIBILITY:
Inclusion Criteria

* Eligible for induction of labor
* Live singleton gestation ≥37 weeks and <42 weeks
* Nulliparous, ≥18 years of age with no previous deliveries >20 weeks
* Cephalic presentation
* Intact membranes
* Bishop score ≤8 and cervical dilation <3 cm
* English or Spanish speaking (Able to read/understand consent and instructions)
* Have reliable transportation to get back to the hospital and have a self-reported safe residence to go home to with the Foley catheter

Exclusion Criteria

* Known oligohydramnios (DVP <2cm)
* Known moderate-severe polyhydramnios (AFI ≥30 at time of delivery)
* Concern regarding fetal status during antenatal testing: At provider discretion, but includes fetal decelerations, biophysical profile ≤6/10
* Vaginal bleeding or concern for/known abruption prior to Foley placement
* Chorioamnionitis
* Any fetal growth restriction
* Preeclampsia with severe features
* Severe chronic hypertension
* Type 1 diabetes or poorly controlled pre-gestational diabetes
* Sickle cell disease
* Major fetal anomaly
* Women on therapeutic anticoagulation
* Decreased fetal movement
* HIV Positive (rationale: HIV positive patients require an IV medication at the start of labor induction which cannot be given as an outpatient. There is universal testing of HIV in the 3rd trimester to verify this exclusion criteria)
* Maternal cardiac disease requiring telemetry monitoring throughout induction/labor course

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2300 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Cesarean Delivery | At delivery
  Incidence of cesarean delivery in women randomized to outpatient cervical ripening with the Foley catheter compared to women undergoing routine inpatient cervical ripening

SECONDARY OUTCOMES:
Maternal morbidity incidence | Within 6 weeks of delivery
  Defined as a composite endpoint consisting of at least one occurrence of the following outcomes: postpartum hemorrhage, blood transfusion, endometritis, wound/laceration breakdown or infection, venous thromboembolis and hospital readmission with 6 weeks
Maternal patient satisfaction as measured by the Hollins Martin Birth Satisfaction scale-Revised (BSS-R) | From time of delivery to discharge from hospital, up to 6 weeks from delivery
  Patient satisfaction as measured by the BSS-R with a possible score of 0-40 with 0 equaling the least birth satisfaction
Neonatal morbidity incidence | Within 6 weeks of delivery
  Defined as a composite endpoint consisting of at least one incidence of the following outcomes: acidemia, respiratory failure/insufficiency, hypoxic-ischemic encephalopathy, treatment for hypoglycemia or suspected sepsis
Maternal patient perception of control | From time of delivery to discharge from hospital, up to 6 weeks from delivery
  Measured by the Labour Agentry Scale (LAS), as 29-item questionnaire with higher values reflecting a higher measure of perceived personal control
Maternal overall length of stay | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Measured by hours from admission to postpartum discharge
Maternal postpartum length of stay | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Measured by hours from delivery to postpartum discharge
Neonatal length of stay | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Length of stay from birth to discharge, measured in hours
NICU admission | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Admission to neonatal intensive care unit
NICU stay greater than 48 hours | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Admission to the NICU for more than 48 hours
Perceived stress scale-10 questions | From time of delivery to discharge from hospital, up to 6 weeks from delivery
  A validated 10 question scale evaluating perceived stress

OTHER OUTCOMES:
Heterogeneity of Treatment Effect/prespecified sub-groups | within 6 weeks of delivery
  Pre-specified subgroups to be included are: Starting cervical dilation (<1cm vs. >=1cm), Bishop score (<6 vs. >=6), BMI (<30 kg/m2 vs. >=30 kg/m2), Race/ethnicity (Black, White, Asian, Other; Hispanic/Non-Hispanic), Gestational age at start of induction (37-39w6d vs. >=40 weeks), Advanced Maternal Age (AMA) (>=35 yo) vs not AMA (<35 yo)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, MD, MSCE, Principal Investigator — University of Pennsylvaina; Alison Cahill, MD, MSCI, Principal Investigator — University of Texas at Austin
Locations (6):
- United States (6):
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Princeton Medical Center, Plainsboro, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - Intermountain Health Utah Valley Hospital, Provo, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: To be determined